CLINICAL TRIAL: NCT00966693
Title: Phase I/II Study of Lenalidomide (Revlimid), Thalidomide, and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Lenalidomide, Thalidomide and Dexamethasone in Treating Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0179; NCI-2018-01857 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0179 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, thalidomide, dexamethasone) (Experimental): Participants receive lenalidomide PO on days 1-21 and thalidomide PO QD on days 1-28. Participants also receive dexamethasone PO QD on days 1-4, 9-12, and 17-20 of courses 1-2, and days 1, 8, 15, and 22 of subsequent courses. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Participants who have stable or responding disease to treatment receive lenalidomide PO on days 1-21 and thalidomide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants may receive dexamethasone at the discretion of the investigator.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide; Drug: Thalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Thalidomide — Given PO
  Other Names: (+)-Thalidomide; (-)-Thalidomide; .alpha.-Phthalimidoglutarimide; 2, 6-Dioxo-3-phthalimidopiperidine; Alpha-Phthalimidoglutarimide; Contergan; Distaval; Kevadon; N-(2,6-Dioxo-3-piperidyl)phthalimide; N-Phthaloylglutamimide; N-Phthalylglutamic Acid Imide; Neurosedyn; Pantosediv; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (+)-; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (-)-; Sedalis; Sedoval K-17; Softenon; Synovir; Talimol; Thalomid

SUMMARY:
This phase I/II trial studies the best dose and side effects of lenalidomide and thalidomide, and how well they work with dexamethasone in treating participants with multiple myeloma that has come back or does not respond to treatment. Drugs used in chemotherapy, such as lenalidomide, thalidomide and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of the combination of lenalidomide and thalidomide and dexamethasone (LTD) in patients with relapsed/refractory multiple myeloma (RRMM). (Phase 1) II. To determine the overall (complete remission [CR)]+ very good partial response [VGPR]+ partial response [PR)] response rate of the combination after 4 cycles of therapy. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR). (Phase 1) II. To determine the time to progression (TTP). (Phase 1) III. To determine the progression free survival (PFS). (Phase 1) IV. To determine the time to best response. (Phase 1) V. To determine the CR, VGPR. (Phase 2) VI. To determine the time to progression (TTP). (Phase 2) VII. To determine the progression free survival (PFS). (Phase 2) VIII. To determine the time to best response. (Phase 2) IX. To assess the safety of the combination of LTD in patients with RRMM. (Phase 2) X. Time to next therapy. (Phase 2) XI. Symptom measurement - multiple-symptom assessment tool. (Phase 2)

OUTLINE: This is a dose-escalation study of lenalidomide and thalidomide.

Participants receive lenalidomide orally (PO) on days 1-21 and thalidomide PO once daily (QD) on days 1-28. Participants also receive dexamethasone PO QD on days 1-4, 9-12, and 17-20 of courses 1-2, and days 1, 8, 15, and 22 of subsequent courses. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Participants who have stable or responding disease to treatment receive lenalidomide PO on days 1-21 and thalidomide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants may receive dexamethasone at the discretion of the investigator.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Relapsed/refractory multiple myeloma (MM) with measurable levels of myeloma paraprotein in serum (>= 0.5 g/dl), urine (>= 0.2 g excreted in a 24-hour collection sample), or abnormal free light chain (FLC) ratio
* Serum creatinine =< 2.5 mg/dl
* Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mlU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Absolute neutrophil count > 1000 cells/mm^3
* Platelet count > 50,000 cells/mm^3 for patients with < 50% of bone marrow plasma cells and platelet count > 25,000 cells/mm^3 for patients in whom > 50% of the bone marrow nucleated cells were plasma cells
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 x upper limit of normal (ULN)
* Able to take prophylactic anticoagulation, warfarin or equivalent agent
* Patient is able to understand and comply with the terms and conditions of the lenalidomide and thalidomide counseling program
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist, AND the S.T.E.P.S. program

Exclusion Criteria:

* Any serious medical condition, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide)
* Use of any cancer therapy within 21 days prior to beginning cycle 1 day 1 of therapy (radiation therapy allowed within 5 days of completion of radiation therapy).
* Known hypersensitivity to thalidomide, lenalidomide and dexamethasone.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-08-25 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Weber, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- RTD (Cohort 1, Phase 1): Oral Revlimid 15mg, Thalidomide 100mg, Dexamethasone 40mg*21 days+ 7 days rest and reevaluation=28 day cycle
- RTD (Cohort 2, Phase 1); RTD (Cohort 2, Phase 2): Oral Revlimid 25mg, Thalidomide 100mg, Dexamethasone 40mg *21 days+ 7 days rest and reevaluation=28 day cycle
- RTD (Cohort 3, Phase 1): Oral Revlimid 25mg, Thalidomide 200mg, Dexamethasone 40mg*21 days+ 7 days rest and reevaluation=28 day cycle
Period: Overall Study
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Started | 3 | 3 | 9 | 49
Phase 1 Completed | 2 | 3 | 6 | 0
Phase 2 Completed | 0 | 0 | 0 | 46
Completed | 2 | 3 | 6 | 26
Not Completed | 1 | 0 | 3 | 23
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 5
Not completed — Disease Progression | 0 | 0 | 1 | 16

BASELINE CHARACTERISTICS:
Groups:
- RTD (Cohort 2, Phase 1); RTD (Cohort 2, Phase 2): Oral Revlimid 25mg, Thalidomide 100mg, Dexamethasone *21 days+ 7 days rest and reevaluation=28 day cycle
- Total: Total of all reporting groups
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2) | Total
Number analyzed (Participants) | 3 | 3 | 9 | 49 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 1 | 26 | 29
  >=65 years | 3 | 1 | 8 | 23 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 19 | 23
  Male | 2 | 3 | 6 | 30 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 3 | 3 | 9 | 46 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 10 | 18
  White | 1 | 1 | 5 | 38 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 9 | 49 | 64
Relapsed/Refractory Multiple Myeloma [Count of Participants; unit: Participants] — Measurable level of disease refractory to previous treatment, study medication tolerance, and able to comply w/ medication regime.
  Participants
    Age >= 18 years old | 3 | 3 | 9 | 49 | 64
    > = 1 line of previous therapy | 3 | 3 | 9 | 49 | 64
    Measurable levels of myeloma >=.5M serum-Protein | 2 | 2 | 7 | 44 | 55
    Measurable levels of myeloma >=.2 Urine-Protein | 0 | 1 | 7 | 42 | 50
    Abnormal Free Light Chain Ratio | 2 | 3 | 9 | 46 | 60
    Creatine < 2.5 mg/dL | 3 | 3 | 9 | 49 | 64
    Platelets > 50,000 | 3 | 3 | 9 | 47 | 62
    Total Bilirubin < 2.0 | 3 | 3 | 9 | 49 | 64
    AST or ALT < 3x Upper Limit | 3 | 3 | 9 | 49 | 64
    Anti-coagulant tolerance (PTT) normal | 2 | 3 | 4 | 37 | 46
    Cognitively Aware & Physically Able | 2 | 2 | 7 | 45 | 56
    No Pregnant/Breast Feeding Females | 1 | 3 | 9 | 19 | 32
    Females non-procreative sex | 1 | 3 | 9 | 19 | 32
    Men non-procreative sex | 2 | 3 | 9 | 30 | 44
    No Cancer Therapy in 21 days | 3 | 3 | 9 | 49 | 64
    No Desquamating Rash regarding Thalidomide | 3 | 3 | 9 | 49 | 64
    Days off prev treatment >= 25 | 3 | 3 | 9 | 44 | 59
    No Known Study Drug Allergies | 3 | 3 | 9 | 49 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limitations Toxicities of the Combination of Lenalidomide and Thalidomide and Dexamethasone (LTD) in Patients With Relapsed/Refractory Multiple Myeloma (RRMM)
Description: To determine the dose limitations toxicities of the combination of lenalidomide and thalidomide and dexamethasone (LTD) in patients with relapsed/refractory multiple myeloma (RRMM).
Time Frame: After one 28-day cycle
Measure: Count of Participants; unit: Participants
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 3 | 3 | 9 | 49
Participants | 1 | 0 | 3 | 0

2. Primary Outcome: Complete Response(CR) and Very Good Partial Response(VGPR)
Description: To determine the best overall response (CR+VGPR+PR) of the lenalidomide, thalidomide, dexamethasone combination based on IMWG criteria at nadir.
Time Frame: Evaluated each 28-day cycle and nadir of criteria is considered best overall response (median time to best response for this study was 2 cycles (range for best overall response was 1-21 cycles).
Measure: Count of Participants; unit: Participants
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 3 | 3 | 9 | 49
Participants
  Partial Remission | 2 | 0 | 2 | 13
  Progressive Disease | 0 | 2 | 2 | 6
  Very Good Partial Remission | 0 | 3 | 1 | 8
  Minimal Residual Disease | 0 | 0 | 1 | 9
  Stringent Complete Remission | 0 | 0 | 0 | 3
  Non Evaluable | 1 | 0 | 3 | 7
  Stable Disease | 0 | 0 | 0 | 7

3. Secondary Outcome: Time to Progression
Description: Time to Progression was estimated using Kaplan Meier analysis.
Time Frame: Up to 9 years
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 3 | 3 | 9 | 49
Months | 32.74 (27) | 9.04 (7.49) | 14.61 (16.41) | 10.02 (17.61)

4. Secondary Outcome: Progression Free Survival
Description: Estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups was made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.
Time Frame: Up to 9 years
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 3 | 3 | 9 | 49
Months | 32.74 (27) | 9.04 (7.49) | 14.61 (16.41) | 10.02 (17.61)

5. Secondary Outcome: Time to Best Response
Description: as for outcome 4
Time Frame: Up to 9 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 3 | 3 | 9 | 49
months | 19 (1.41) | 5 (6.08) | 5.16 (7.03) | 3.3 (4.2)

6. Secondary Outcome: Incidence of Adverse Events
Description: Linear regression was utilized to assess the effect of patient prognostic factors on the toxicity rate.
Time Frame: Up to 9 years
Population: The Number in each of the arms was insufficient to conduct regression analyses, therefore regression analyses was conducted overall. Participants who were Thalidomide incompatible.
Measure: Count of Participants; unit: Participants
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 2 | 3 | 6 | 49
Participants | 0 | 0 | 2 | 10

7. Secondary Outcome: Time to Next Therapy
Description: Estimated using the method of Kaplan and Meier.
Time Frame: Up to 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
Number analyzed (Participants) | 3 | 3 | 9 | 49
months | 52.4 [1.94 to NA] — insufficient number of participants with events | 14.3 [5.19 to NA] — insufficient number of participants with events | 10.5 [4.96 to NA] — insufficient number of participants with events | 6.47 [4.14 to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Baseline to study completion up to 9 years
Arm/Group | RTD (Cohort 1, Phase 1) | RTD (Cohort 2, Phase 1) | RTD (Cohort 3, Phase 1) | RTD (Cohort 2, Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/9 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/9 | 7/49
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 9/9 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTD (Cohort 1, Phase 1) (N=3) | RTD (Cohort 2, Phase 1) (N=3) | RTD (Cohort 3, Phase 1) (N=9) | RTD (Cohort 2, Phase 2) (N=49)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 1
Altered Mental Status (Psychiatric disorders) | 0 | 0 | 0 | 2
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTD (Cohort 1, Phase 1) (N=3) | RTD (Cohort 2, Phase 1) (N=3) | RTD (Cohort 3, Phase 1) (N=9) | RTD (Cohort 2, Phase 2) (N=49)
Activated PTT (Investigations) | 1 | 3 | 7 | 12
Acidosis (Investigations) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Adult Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
ALT Increase (Investigations) | 2 | 1 | 5 | 16
Alkaline Phosphate increase (Investigations) | 1 | 1 | 4 | 7
Allergy (Immune system disorders) | 0 | 1 | 1 | 1
Anal Hemmorhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 5
Anxiety (Psychiatric disorders) | 1 | 0 | 3 | 8
AST Increase (Investigations) | 2 | 1 | 4 | 19
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 2 | 4
Atrial Injury (Cardiac disorders) | 0 | 0 | 0 | 1
Auditory Ear (Other) (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Autoimmune Disorder (Other) (Immune system disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 20
Hyperbilirubia (Investigations) | 1 | 0 | 3 | 10
Hypocarpnia (Investigations) | 0 | 0 | 0 | 2
Hyperglycemia (Investigations) | 2 | 3 | 7 | 45
Hyperuricemia (Investigations) | 1 | 2 | 1 | 18
Blood Bone Marrow (other) (Investigations) | 0 | 0 | 0 | 1
Bone Development Abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
BonePain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Bronchial Hemmorhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Brusing (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Cardiac General (Other) (Cardiac disorders) | 0 | 1 | 1 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 1
Hypocaligulopathy (Investigations) | 1 | 3 | 6 | 7
Confusion (Psychiatric disorders) | 0 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 2 | 1 | 6 | 33
Conjunctival disorder (Eye disorders) | 0 | 0 | 0 | 1
Constitutional Symptoms (General disorders) | 1 | 0 | 0 | 2
Cushingoid (Endocrine disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 17
Creatinine increase (Investigations) | 1 | 0 | 5 | 27
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Dehydration (General disorders) | 0 | 0 | 0 | 5
Depressed Conciousness Level (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3
Dermatological/Skin (other) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 5 | 32
Diastolic Dysfunction (Cardiac disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 6 | 31
Dry Eye Syndrome (Eye disorders) | 1 | 0 | 1 | 20
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7 | 38
Edema Limbs (General disorders) | 2 | 3 | 8 | 36
Endocrine (other) (Endocrine disorders) | 0 | 0 | 0 | 1
Esophogeal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Eye Muscle Weakness (Eye disorders) | 0 | 0 | 0 | 1
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 9 | 49
Fever (General disorders) | 2 | 1 | 2 | 17
Flashing Vision (Eye disorders) | 0 | 0 | 1 | 0
Flu-like Symptoms (General disorders) | 0 | 0 | 1 | 2
Gait Abnormal (Nervous system disorders) | 0 | 0 | 0 | 1
Gastric Infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal General (Gastrointestinal disorders) | 1 | 0 | 2 | 7
Glucose intolerance (Endocrine disorders) | 0 | 1 | 0 | 1
Headache (General disorders) | 0 | 1 | 0 | 10
Hearing Loss (Ear and labyrinth disorders) | 1 | 0 | 1 | 1
Hematoma (Vascular disorders) | 0 | 0 | 2 | 2
Anemia (Investigations) | 3 | 1 | 6 | 43
Epstaxis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hemorrhoidal/hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhage Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hiccough (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypercalcemia (Investigations) | 0 | 0 | 0 | 10
Hypertension (Cardiac disorders) | 0 | 0 | 1 | 5
Hypotension (Cardiac disorders) | 1 | 0 | 1 | 8
Infection (Infections and infestations) | 1 | 1 | 2 | 11
INR Increase (Investigations) | 1 | 1 | 3 | 7
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 8
Irratibility (Psychiatric disorders) | 0 | 0 | 1 | 1
Jejunal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Joint Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Leukopenia (Investigations) | 2 | 2 | 6 | 35
Lymphatics (Other) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4
Localized Edema (General disorders) | 1 | 1 | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 13
Memory Impairement (Nervous system disorders) | 2 | 1 | 5 | 30
Metabolic/Laboratory (Other) (Investigations) | 2 | 1 | 8 | 29
Mucosal Infection (Infections and infestations) | 0 | 1 | 1 | 1
Mucositis Oral (Gastrointestinal disorders) | 1 | 1 | 2 | 24
Musculoskeletal (Other) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 12
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1
Musculoskelatal (Other) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7
Myalgia (Nervous system disorders) | 2 | 2 | 2 | 19
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Mycardial Ichemia (Cardiac disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 25
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neurology (Other) (Nervous system disorders) | 2 | 0 | 6 | 10
ANC Decrease (Investigations) | 3 | 0 | 4 | 33
Ocular/Visual (Other) (Eye disorders) | 2 | 0 | 2 | 3
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Osteoporsis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Otitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Pain (Nervous system disorders) | 0 | 0 | 3 | 30
Pain (Other) (Nervous system disorders) | 0 | 0 | 2 | 4
Pain in extremity (Nervous system disorders) | 1 | 1 | 2 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 7 | 41
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pharyngitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Photosensitivity (Eye disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Thromboctopenia (Investigations) | 2 | 1 | 6 | 30
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 13
Proteinuria (Investigations) | 0 | 1 | 1 | 3
Pulmonary (Other) (Cardiac disorders) | 1 | 0 | 0 | 7
Rash acneform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Renal/Genitourinary (Other) (Renal and urinary disorders) | 1 | 0 | 0 | 3
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Hypoalbumenia (Investigations) | 2 | 2 | 9 | 33
Hypocalcemia (Investigations) | 1 | 2 | 8 | 25
Hypomagnesemia (Investigations) | 1 | 1 | 4 | 33
Hypermagnesmia (Investigations) | 0 | 0 | 1 | 0
Hypoglycemia (Investigations) | 0 | 0 | 1 | 4
Hypophosphatemia (Investigations) | 1 | 1 | 4 | 17
Hyperkalemia (Investigations) | 1 | 0 | 1 | 17
Hypokalemia (Investigations) | 1 | 0 | 3 | 11
Hyponatremia (Investigations) | 2 | 1 | 4 | 11
Hypernatremia (Investigations) | 0 | 0 | 1 | 3
Hypercholesteremia (Investigations) | 0 | 0 | 0 | 1
Sinus Brdaycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 4
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 2
Hyperhidrosis (General disorders) | 0 | 0 | 0 | 3
Taste Alteration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tinitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Speech Disorder (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Treatment related to Secondary Malignancy (Surgical and medical procedures) | 0 | 0 | 0 | 4
Tremor (Nervous system disorders) | 0 | 0 | 2 | 8
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 18
Urinary Urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 0 | 0 | 2 | 9
Urostomy stenosis (Surgical and medical procedures) | 0 | 0 | 0 | 1
Vaginal hemmorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 2 | 1 | 7 | 29
Vascular (other) (Vascular disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 16
Voice Alteration (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Watering Eyes (Eye disorders) | 2 | 1 | 1 | 21
Weight Gain (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3

LIMITATIONS AND CAVEATS:
No pharmaco-dynamic marker to support an effect of signaling downregulation in lenalidomide-refractory patients to corroborate low dose thalidomide (50-100 mg) with or without dexamethasone has a therapeutic benefit with lenalidomide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT00966693/Prot_SAP_000.pdf